CLINICAL TRIAL: NCT02877693
Title: A Post-market Clinical Evaluation of St. Jude Medical™ MR Conditional ICD System on Patients Undergoing Magnetic Resonance Imaging
Acronym: ASIA MRI ICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SJM-CIP-10163
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Results first posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-03

CONDITIONS: ICD; Tachycardia
Keywords: ICD; Thoracic MRI Scan; tachycardia
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thoracic MRI Scan with 1.5 Tesla MRI (Experimental): Subjects will be enrolled at least 60 days post successful St. Jude Medical™ MR Conditional ICD System implant. Enrolled subjects will undergo an elective 1.5T MRI scan within 30 days post enrollment. Post MRI visit all subjects will be followed up at 1-Month post MRI visit.
  Interventions: Radiation: Thoracic MRI Scan
- Thoracic MRI Scan with 3 Tesla MRI (Experimental): Subjects will be enrolled at least 60 days post successful St. Jude Medical™ MR Conditional ICD System implant. Enrolled subjects will undergo an elective 3T MRI scan within 30 days post enrollment. Post MRI visit all subjects will be followed up at 1-Month post MRI visit.
  Interventions: Radiation: Thoracic MRI Scan

INTERVENTIONS:
Radiation: Thoracic MRI Scan — The ICD system will be exposed to MRI scan of thoracic region, where the radiofrequency (RF) component of the scan is maximized.

SUMMARY:
To assess the clinical performance of the St. Jude Medical™ MR Conditional ICD System in patients undergoing an elective thoracic MRI scan.

DETAILED DESCRIPTION:
This clinical investigation is a prospective, multicenter, Asian study. The study was designed with two (2) parts, however only the 1st part was completed. For the 1st part, patients were enrolled with a SJM MR Conditional ICD System approved for thoracic scan with 1.5 Tesla MRI scanning machines. The 2nd part-meant to enroll patients for thoracic scans with 3 Tesla MRI scanning machines-was not completed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is pectorally implanted with St. Jude Medical™ MR Conditional ICD System for at least 60 days
2. Subject is willing to undergo an elective MRI scan without sedation NOTE: Antianxiety agents (e.g. minor tranquilizers, etc.) may be used as long as the patient can communicate with site personnel during the MRI scan
3. Subject's ventricular bipolar capture threshold is stable < 2.5V @ 0.5ms
4. Subject's ventricular sensing is measurable (patient has underlying rhythm > 30bpm) and the sensing amplitude is stable > 4mV
5. Subject is able to provide informed consent for study participation (legal guardian or legally authorized representative is NOT acceptable)
6. Subject is willing and able to comply with the prescribed follow-up tests and procedures
7. Subject is not contraindicated for an MRI scan (per the MRI Screening Form)

Exclusion Criteria:

1. Subject is pacemaker dependent
2. Subject has a non SJM MRI compatible endocardial lead implanted or capped
3. Subject has another existing active implanted medical device, e.g., neurostimulator, infusion pump, etc. that has MR labeling that will not allow the MRI scans per this protocol to be completed.
4. Subject has a high voltage lead revision incidence < 60 days of the enrollment visit
5. Subject has other non-MRI compatible device or material implanted NOTE: MRI compatible knee replacements, hip replacements, stents, etc. may be included as long as the labeling of these devices allow MRI scans conducted per this protocol NOTE: MRI compatible mechanical, prosthetic, and bioprosthetic heart valves may be included as long as the labeling of these devices allow for MRI scans conducted per this protocol NOTE: Non-removable dental implants may be included
6. Subject has a lead extender, adaptor, or capped/abandoned lead
7. Subject is enrolled or intend to participate in a clinical drug and/or device study (investigational device, investigational drug, new indication for a device or drug or additional testing beyond standard of care procedures), which could confound the results of this trial as determined by SJM.
8. Subject is pregnant or planning to become pregnant during the duration of the subject's participation in the study
9. Subject has a life expectancy of less than 12 months due to any condition
10. Subject has exclusion criteria required by local law (e.g., age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant Kim, Study Director — St. Jude Medical, Inc.
Locations (20):
- India (14):
  - Medanta-The Medicity, Gurgaon, Haryana
  - Post Graduate Institute of Medical Education & Research, Chandigarh
  - BLK Super Speciality Hospital, Delhi
  - Max Super Specialty Hospital, Delhi
  - Pushpawati Singhania Research Institute, Delhi
  - Apollo Gleneagles Hospital, Delhi
  - Batra Hospital & Medical Research Centre, Delhi
  - Fortis Flt. Lt. Rajan Dhall Hospital, Delhi
  - National Heart Institute, Delhi
  - Medanta Medicity Hospital, Gūrgaon
  - Care Hospital, Hyderabad
  - Asian Heart Institute, Mumbai
  - Escorts Heart Institute and Research Centre, New Delhi
  - Ruby Hall Clinic, Pune
- Hospital Serdang, Kajang, Malaysia
- South Korea (5):
  - Dankook University Hospital, Cheonan
  - Cha Bundang Medical Center, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tarlochan Singh Kler, Praveen Chandra, Chandrakant Chavan, Rajesh Vijayvergiya, Subhash Chandra, Anoop Gupta, Sridevi Chennapragada, Joung Bo Young, Mona Bhatia, Choi Eue Keun, Vanita Arora, Tom Devasia, Upendra Kaul, Sumit Anand, Kartikeya Bhargava. Initial experience of thoracic Magnetic Resonance Imaging (MRI) scanning in Asian patients implanted the Ellipse MR Conditional ICD System - The ASIA MRI ICD Study. APHRS 2017; Abstract no. 40528.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject enrollment in the Asia MRI ICD study began on October 10, 2016. The study enrolled 205 subjects at 20 clinical sites. Completion of enrollment and follow-up in the study occurred on March 23, 2020.
Period: Overall Study
Arm/Group | Thoracic MRI Scan With 1.5 Tesla MRI | Thoracic MRI Scan With 3 Tesla MRI
Started | 205 | 0 (This arm was not completed. As of the data cut-off date for this clinical study report subject enrollment criteria was met for the 1st arm of the study and the sponsor decided not to move forward with 3T arm of the study.)
Completed | 177 | 0
Not Completed | 28 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consisted of study participants that provided and signed acknowledgement of informed consent and were enrolled in the study.
Arm/Group | Thoracic MRI Scan With 1.5 Tesla MRI
Number analyzed (Participants) | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 178
  Unknown or Not Reported | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 201
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  South Korea | 20
  Malaysia | 4
  India | 181
Cardiovascular History [Count of Participants; unit: Participants]
  Non-ischemic Cardiomyopathy | 75
  Ischemic Cardiomyopathy | 93
  No Cardiomyopathy | 37
Primary Indication for ICD Implant [Count of Participants; unit: Participants]
  Cardiac Arrest | 22
  Ventricular Tachycardia | 57
  Ischemic Cardiomyopathy | 61
  Non-ischemic Cardiomyopathy | 50
  Syncope | 9
  Familial Condition | 2
  Other | 4
History of Smoking [Count of Participants; unit: Participants]
  Number of years smoking < 10 | 9
  Number of years smoking 10 - 20 | 8
  Number of years smoking > 20 | 12
  No smoking or no response | 176

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Freedom From MRI-scan Related Complications* Related to St. Jude Medical™ MR Conditional ICD System
Description: *A complication is a serious adverse device effect (SADE) that requires an invasive intervention or leads to death.
  The primary endpoint analysis will be performed for each study phase separately.
Time Frame: from MRI scan visit to 1 month post-MRI scan visit
Population: 177 subjects (86.3% of enrolled subjects) completed through the 1-month post-MRI scan visit and are included in the primary safety endpoint analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic MRI Scan With 1.5 Tesla MRI
Number analyzed (Participants) | 177
Participants | 177

2. Other Pre Specified Outcome: The Average Specific Absorption Rate (SAR)
Description: The average Specific Absorption Rate (SAR) during the MRI scan
Time Frame: MRI scan visit
Population: Subjects completing the MRI scan in its entirety
Measure: Mean (Standard Deviation); unit: Watts/kg
Arm/Group | Thoracic MRI Scan With 1.5 Tesla MRI
Number analyzed (Participants) | 180
Watts/kg | 1.9 (0.2)

3. Other Pre Specified Outcome: Number of Participants With Freedom From MRI-scan Related Complications* Related to St. Jude Medical™ MR Conditional ICD System
Description: This proportion was calculated as the number of subjects who had high voltage leads with capture threshold increases of ≤ 0.5V @ 0.5 ms from pre MRI scan testing to 1-month post MRI scan testing divided by total number of subjects who had high voltage lead implanted, underwent an MRI scan and had both pre-MRI scan and 1-month post MRI scan capture threshold measurements available.
Time Frame: from MRI scan visit to 1-month post MRI scan visit
Population: Subjects who had high voltage lead implanted, underwent an MRI scan and had both pre MRI scan and 1 month post MRI scan sensing amplitudes available
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic MRI Scan With 1.5 Tesla MRI
Number analyzed (Participants) | 172
Participants | 168

4. Other Pre Specified Outcome: Proportion of SJM High Voltage Lead Implanted With SJM MR Conditional ICD With Sensing Amplitude Decrease of ≤ 50% From Pre-MRI Scan Testing to 1 Month Post-MRI Scan Testing
Description: This proportion was calculated as the number of subjects who had high voltage leads with sensing amplitude decrease of ≤ 50% from pre MRI scan testing to 1 month post MRI scan testing divided by the total number of subjects who had high voltage lead implanted, underwent an MRI scan and had both pre MRI scan and 1 month post MRI scan sensing amplitudes available.
Time Frame: from pre MRI scan to 1-month post MRI scan
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic MRI Scan With 1.5 Tesla MRI
Number analyzed (Participants) | 174
Participants | 173

5. Other Pre Specified Outcome: The Peak Specific Absorption Rate (SAR) During the MRI Scan
Description: The peak Specific Absorption Rate (SAR) during the MRI scan
Time Frame: MRI Scan Visit
Population: The peak SAR was calculated for 56 subjects with available data
Measure: Mean (Standard Deviation); unit: W/kg
Arm/Group | Thoracic MRI Scan With 1.5 Tesla MRI
Number analyzed (Participants) | 56
W/kg | 1.5 (0.3)

6. Other Pre Specified Outcome: The Mean MRI Visit Duration in the MRI Lab
Description: The mean MRI visit duration in the MRI lab
Time Frame: MRI Visit
Population: The mean MRI visit duration in the MRI lab for 181 subjects completing the MRI scan visit
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Thoracic MRI Scan With 1.5 Tesla MRI
Number analyzed (Participants) | 181
minutes | 37.3 (11.1)

7. Other Pre Specified Outcome: Total MRI Scan Duration in MRI Laboratory
Description: Total MRI scan duration in MRI laboratory
Time Frame: MRI Visit
Population: Subjects completing the MRI scan
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Thoracic MRI Scan With 1.5 Tesla MRI
Number analyzed (Participants) | 180
minutes | 24.4 (1.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time participants were enrolled, through the MRI scan Visit and the 1 month Post MRI Scan Visit follow-up, or the study completion (if subject withdrawn before the final follow-up).
Description: * Adverse Device Effect (ADE)- An adverse event (AE) related to the use of a medical device. This definition includes AEs resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the medical device and any event resulting from the use error or from intentional misuse of the medical device.
  * Serious Adverse Device Effect - ADE that has resulted in any of the consequences characteristic of a Serious AE
Arm/Group | Thoracic MRI Scan With 1.5 Tesla MRI
All-Cause Mortality (participants affected / at risk) | 2/205
Serious Adverse Events (participants affected / at risk) | 1/205
Other Adverse Events (participants affected / at risk) | 1/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thoracic MRI Scan With 1.5 Tesla MRI (N=205)
Breathlessness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Refractory cardiogenic shock, recurrent ventricular tachycardia, ventricular fibrillation (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Serious Adverse Device Effect: Acute Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — *Event was conservatively classified as SADE due to unknown relationship to the device per the investigator's assessment.
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thoracic MRI Scan With 1.5 Tesla MRI (N=205)
Loss of Capture (Product Issues) | 1 (1) — Device loss of capture

LIMITATIONS AND CAVEATS:
The 3T MRI part of the study was not completed as the study was terminated upon completion of the 1.5T MRI part of the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT02877693/Prot_SAP_000.pdf